CLINICAL TRIAL: NCT07314853
Title: Fluid Optimization in Cancer Surgery With AI-Assisted Management - FOCUS-AFM Trial
Brief Title: Using Artificial Intelligence to Guide Fluid Therapy During Major Cancer Surgery: A Randomized Controlled Trial
Acronym: FOCUS-AFM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOCUS AFM
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Neoplasm; Cancer; Hemodynamic (MAP) Stability; Cancer Surgery; Artificial Intelligence (AI); Fluid Therapy DURING SURGERY
Keywords: randomized controlled trial; cancer; fluid balance; fluid therapy; artificial intelligence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Fluid Management (Active Comparator): Participants receive intraoperative intravenous fluid therapy managed according to usual clinical practice, without artificial intelligence guidance. Fluid administration is determined by the attending clinician based on standard monitoring and clinical judgment.
  Interventions: Other: Standard fluid management
- AI-Assisted Fluid Management (Experimental): Participants assigned to this arm receive intraoperative intravenous fluid therapy supported by an artificial intelligence-based clinical decision support system. The system analyzes real-time hemodynamic data and provides recommendations for fluid administration. Clinicians are strongly encouraged to follow these recommendations but may accept or override them based on clinical judgment.
  Interventions: Other: Artificial Intelligence-Assisted Fluid Management

INTERVENTIONS:
Other: Artificial Intelligence-Assisted Fluid Management — In this intervention, intraoperative intravenous fluid management is supported by an artificial intelligence-based clinical decision support system. The system continuously analyzes real-time hemodynamic data derived from standard intraoperative monitoring and provides recommendations for intravenous fluid administration. Clinicians are strongly encouraged to follow these recommendations but retain full responsibility and may accept or override them based on clinical judgment. The intervention is applied during the intraoperative period only and does not replace standard anesthetic care.
  Arms: AI-Assisted Fluid Management
Other: Standard fluid management — In this intervention participants receive intraoperative intravenous fluid therapy managed according to usual clinical practice, without artificial intelligence guidance. Fluid administration is determined by the attending clinician based on standard monitoring and clinical judgment.
  Arms: Standard Fluid Management

SUMMARY:
The goal of this clinical trial is to learn if using artificial intelligence to guide intravenous fluid therapy during major cancer surgery can help keep blood pressure more stable compared with usual care in adult patients undergoing major cancer surgery. The main questions it aims to answer are:

* Does artificial intelligence-guided fluid therapy reduce hypotensive events during surgery?
* Does this approach improve recovery and reduce complications after major cancer surgery?

Researchers will compare artificial intelligence-guided fluid therapy with standard fluid management to see if the artificial intelligence-guided approach provides better support during surgery.

Participants will:

* Undergo major cancer surgery under general anesthesia
* Receive either artificial intelligence-guided fluid management or standard fluid management during surgery
* Be monitored during and after surgery as part of routine clinical care
* Be followed after surgery to assess recovery and possible complications

DETAILED DESCRIPTION:
This multicentre randomized controlled clinical trial evaluates the impact of artificial intelligence-guided intraoperative intravenous fluid therapy on hemodynamic management and postoperative outcomes in adult patients undergoing major abdominal cancer surgery.

Optimal intraoperative fluid therapy is a critical component of anesthetic management during major oncologic surgery. Both inadequate and excessive fluid administration may contribute to hemodynamic instability and postoperative complications. Episodes of intraoperative hypotension have been consistently associated with increased postoperative morbidi ty and mortality, particularly in high-risk surgical populations. Although goal-directed strategies for intraoperative fluid therapy have been proposed, their implementation in routine clinical practice remains heterogeneous and highly operator-dependent.

Advances in artificial intelligence have enabled the development of decision support systems capable of integrating continuous hemodynamic data derived from standard intraoperative monitoring. These systems are designed to assist clinicians by analyzing multiple physiologic variables in real time and providing recommendations for intravenous fluid administration aimed at supporting circulatory stability, while preserving full clinician control over treatment decisions.

In this trial, participants undergoing major abdominal cancer surgery under general anesthesia are randomly assigned to receive either artificial intelligence-guided intravenous fluid therapy or standard intravenous fluid management according to routine clinical practice. Randomization is centralized and stratified by relevant procedural factors. In the intervention group, intravenous fluid administration is supported by an artificial intelligence-based decision support system that continuously analyzes intraoperative hemodynamic data and generates recommendations for fluid challenges. Clinicians are strongly encouraged to follow the system recommendations; however, they retain full responsibility and may accept or override these recommendations based on their clinical judgment. In the control group, intraoperative fluid therapy is managed according to usual clinical practice without artificial intelligence guidance.

Standard perioperative monitoring is applied in both study groups, including continuous invasive arterial blood pressure monitoring. Intraoperative hemodynamic variables, fluid administration, and use of vasoactive medications are recorded prospectively using electronic anesthesia records and monitoring system outputs. Postoperative clinical data are collected during routine inpatient care and scheduled follow-up.

The study focuses on the intraoperative period as a key window during which hemodynamic management may influence postoperative recovery and longer-term outcomes. By evaluating an artificial intelligence-based decision support approach in a randomized multicentre setting, this trial aims to generate evidence on whether technology-assisted intravenous fluid therapy can improve intraoperative management and support better clinical outcomes in patients undergoing major cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) Physical Status II-IV
* Undergoing major abdominal oncologic surgery (open or laparoscopic) with an expected duration >2 hours
* Planned invasive arterial pressure monitoring
* Ability to understand and sign informed consent

Exclusion Criteria:

* Significant arrhythmias (e.g., persistent atrial fibrillation)
* Severe aortic stenosis
* Emergency surgery
* Sepsis
* End-stage renal disease on dialysis
* Pregnancy
* Impossibility to cannulate the radial artery
* Refusal to participate or refusal of data processing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Hypotension Burden | From induction of anesthesia to the end of surgery
  The burden of intraoperative hypotension, measured as the time-weighted average (TWA) of intraoperative hypotension, a composite measure that accounts for both the depth and duration of low arterial blood pressure over time. TWA reflects the overall hypotensive burden during surgery by integrating how low blood pressure falls and for how long it remains below predefined thresholds, assessed using continuous invasive blood pressure monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Nazionale Tumori "Fondazione G. Pascale", Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes